CLINICAL TRIAL: NCT05271097
Title: Developing a MHealth HIV Prevention Intervention for Transgender Women (Phase 1 and 2)
Brief Title: MHealth HIV Prevention for Transgender Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000030146; 1R21AI157857-01A1 (NIH)
Record Dates: First submitted 2022-02-24; First posted 2022-03-08 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: HIV
Keywords: transgender; HIV prevention; HIV intervention; transgender woman

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MyLink2Care app (Experimental): Participants in the MyLink2Care group will be provided with full app access and will be encouraged to use all features of the app.
  Interventions: Other: MyLink2Care app full functionality
- treatment-as-usual (TAU) (Active Comparator): Participants in the TAU group will receive the MyLink2Care app with major intervention features inactivated.
  Interventions: Other: MyLink2Care app major intervention features inactivated

INTERVENTIONS:
Other: MyLink2Care app full functionality — Participants will be shown how to download the app and use the assessment tool.
  Arms: MyLink2Care app
Other: MyLink2Care app major intervention features inactivated — Participants will be shown how to download the app and use the assessment tool.
  Arms: treatment-as-usual (TAU)

SUMMARY:
This study aims to inform the development of an acceptable and usable smartphone app for transgender women (TGW) in Malaysia to deliver an integrated HIV prevention intervention that incorporates screening and guidance for HIV testing and pre-exposure prophylaxis compared to treatment as usual.

DETAILED DESCRIPTION:
This study aims to inform the development of an acceptable and usable smartphone app for transgender women (TGW) in Malaysia to deliver an integrated HIV prevention intervention that incorporates screening and guidance for HIV testing and pre-exposure prophylaxis (PrEP) compared to treatment as usual.

A new clinic-affiliated app (to be called MyLink2Care) will be developed (by adapting an existing app) and tested to deliver an integrated HIV prevention intervention that incorporates tailored HIV prevention and gender affirming care (GAC) services to TGW in Malaysia. The specific aims of the study include:

* Aim 1: Guided by the modified IM Adapt model, an existing mobile app will be adapted, expanded, and refined. Focus groups will be conducted with TGW (n=20) and clinical stakeholders (n=10) to theater test the existing app to develop an interactive prototype of the MyLink2Care app (alpha version), which will undergo usability testing (N=10), followed by full development of the app (beta version).
* Aim 2 Conduct beta testing of the fully developed version of the MyLink2Care app (N=15) to assess its usability and acceptability.
* Aim 3: Assess preliminary feasibility and acceptability of the MyLink2Care app within a pilot, randomized controlled trial, compared with treatment as usual for engagement in the HIV prevention cascade (N=50).

Together, these aims will address multilevel barriers to HIV testing and PrEP uptake in Malaysian TGW. Feasibility is high based on the investigators extensive experience with HIV prevention in TGW, theory-guided behavioral interventions, mHealth expertise, and longstanding work in Malaysia.

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative
* Identify as a transgender woman
* Condomless sex in the last 30 days
* Own a smartphone

Exclusion Criteria:

* Unable to provide informed consent
* Unable to read and understand English or Bahasa Malaysia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender women
Enrollment: 50 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the MyLink2Care app using percentages of individuals screened | 6 months
  The investigators will use the percentage of individuals screened to determine the feasibility of the MyLink2Care app
Feasibility of the MyLink2Care app using percentages of individuals eligible | 6 months
  The investigators will use the percentage of individuals eligible to determine the feasibility of the MyLink2Care app
Feasibility of the MyLink2Care app using percentages of individuals enrolled | 6 months
  The investigators will use the percentage of individuals enrolled to determine the feasibility of the MyLink2Care app
Feasibility of the MyLink2Care app using percentages of individuals retained | 6 months
  The investigators will use the percentage of individuals retained to determine the feasibility of the MyLink2Care app
Feasibility of the MyLink2Care app using the percentage of participants that accessed the app | 6 months
  The investigators will determine the percentage of participants that accessed the app, with ≥60% of participants accessing app as lower threshold. The higher the percentage, the higher the feasibility.
Acceptability of the MyLink2Care app based on the subjective usability measure | 6 months
  Acceptability will be based on descriptive statistics from the subjective usability measure, with a target mean score of ≥ 50. The higher the score, the higher the acceptability. Minimum score for the scale is 0, highest is 100.
Acceptability of the MyLink2Care app based on perceived usefulness of participants assessed in qualitative interviews | 6 months
  Acceptability will be based on analysis of qualitative data which includes specific areas of perceived usefulness of the app.
Acceptability of the MyLink2Care app based on barriers and facilitators identifies by participants in qualitative interviews | 6 months
  Acceptability will be based on analysis of qualitative data which includes barriers and facilitators
Acceptability of the MyLink2Care app based on usability concerns identified by participants in qualitative interviews | 6 months
  Acceptability will be based on analysis of qualitative data which includes usability concerns.
Acceptability of the MyLink2Care app based on refinement feedback identified by participants in qualitative data interviews | 6 months
  Acceptability will be based on analysis of qualitative data which includes refinement needed to maximize future implementation.

SECONDARY OUTCOMES:
Preliminary Efficacy of the MyLink2Care app through dried blood spot (DBS) testing as PrEP adherence measure | 3 months
  The investigators will measure PrEP adherence DBS at 3 months. DBS will quantify tenofovir-diphosphate (TFV-DP) and emtricitabine-triphosphate (FTC-TP) in red blood cells (RBC).
Preliminary Efficacy of the MyLink2Care app through DBS testing as PrEP adherence measure | 6 months
  The investigators will measure PrEP adherence DBS at 6 months. DBS will quantify tenofovir-diphosphate (TFV-DP) and emtricitabine-triphosphate (FTC-TP) in RBC
Preliminary Efficacy of the MyLink2Care app using the visual analog scale (VAS) to measure PrEP adherence | 3 months
  The investigators will measure PrEP adherence using the visual analogue scale at 3 months
Preliminary Efficacy of the MyLink2Care app using the visual analog scale (VAS) to measure PrEP adherence | 6 months
  The investigators will measure PrEP adherence using the visual analogue scale at 6 months.
Preliminary Efficacy of the MyLink2Care app using proportion of participants who persist on PrEP | 6 months
  Preliminary Efficacy of the app will be calculated using the proportion of participants who persist on PrEP. Persistence on PrEP is measured on the app when completing PrEP care.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Wickersham, PhD, Principal Investigator — Yale University
Locations (1):
- University of Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No